CLINICAL TRIAL: NCT06546397
Title: Prospective Cohort Study on the Effect of Combined Estrogen and Progestogen Therapy on Endometrial Repair and Ovarian Function Recovery After Induced Abortion
Brief Title: Study on the Effect of Combined Estrogen and Progestogen Therapy on Endometrial Repair After Induced Abortion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO2023-3733; BJ2023YCPYJH003 (Other Grant/Funding Number: China Health & Medical Development Foundation)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Complications
Keywords: induced abortion; Intrauterine adhesion; estrogen; endometrial repair
MeSH Terms: conditions — Pregnancy Complications; Gynatresia | interventions — Estradiol; Dydrogesterone

STUDY DESIGN:
Intervention Model Description: The eligible population who underwent induced abortion were divided into two groups using block randomization. The experimental group received estrogen and progesterone therapy after surgery, while the other group served as a blank control group. Twenty-one days after surgery, a follow-up examination was conducted to assess the recovery of the endometrium and measure the endometrial thickness. Twenty-one days after the first post-operative menstrual cycle, blood samples were taken for laboratory tests to evaluate the recovery of ovarian function.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoston group (Experimental): Starting from the day of the induced abortion surgery, take 17β-estradiol/dydrogesterone tablets orally for 28 days (take 2mg of 17β-estradiol orally once a day for the first 14 days, and then take 2mg of 17β-estradiol + 10mg of dydrogesterone tablets orally once a day for the next 14 days).The medication product name is called Femoston。
  Interventions: Drug: 17β-estradiol/dydrogesterone tablets
- No Femoston group (No Intervention): The blank control group did not receive Femoston（17β-estradiol/dydrogesterone tablets after induced abortion surgery.

INTERVENTIONS:
Drug: 17β-estradiol/dydrogesterone tablets — The medication group began taking 17β-estradiol/dydrogesterone tablets orally for 28 days starting from the first day after induced abortion surgery (taking 2mg of 17β-estradiol orally once a day for the first 14 days, and then taking 2mg of 17β-estradiol + 10mg of dydrogesterone tablets orally once a day for the next 14 days). The blank control group did not take any medication.
  Arms: Femoston group

SUMMARY:
Induced abortion is a common method to terminate pregnancy, but during the operation, it is necessary to dilate the cervix and aspirate the uterine cavity. Repeated induced abortions may increase the risk of uterine damage, leading to cervical stenosis or intrauterine adhesions, thinning of the endometrium, which may affect the implantation of fertilized eggs and the development of embryos, and ultimately may lead to infertility or miscarriage. This study aims to explore the effects of combined estrogen and progesterone on endometrial repair and ovarian function recovery after induced abortion.

DETAILED DESCRIPTION:
Postoperative care after induced abortion should prioritize the issue of endometrial repair. In 2021, the Family Planning Branch of the Chinese Medical Association published the "Expert Consensus on Promoting Endometrial Repair After Induced Abortion" [10], emphasizing the importance of endometrial repair for high-risk populations following induced abortion. Currently, clinically, methods to promote endometrial repair include estrogen-progestin medications, compound short-acting oral contraceptives, traditional Chinese medicine, and bioelectric stimulation. However, controversies still exist regarding endometrial repair, and selecting an effective and safe treatment plan remains crucial. This study aims to prospectively evaluate the efficacy and safety of estradiol/estradiol/dydrogesterone in endometrial repair after induced abortion through clinical research, providing a basis for endometrial repair and ovarian function recovery post-abortion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years old (inclusive) and 40 years old (inclusive)
* Body Mass Index (BMI) ranging from 18.5Kg/㎡ to 23.9Kg/㎡
* Experienced at least 2 abortions or had a missed abortion
* Confirmed gestational age of no more than 10 weeks, and the ultrasonic examination within three days prior to the surgery shows a gestational sac (average of three diameters) of at least 1.0cm, with an embryo length of no more than 3.0cm
* Normal preoperative examination results as per the "Clinical Diagnosis and Treatment Guidelines and Technical Operation Standards: Family Planning Volume (2017 Revision)"
* Capable of regular follow-ups and willing to sign the informed consent form.

Exclusion Criteria:

* Individuals with contraindications to estrogen and progesterone therapy
* History of uterine adhesions confirmed by hysteroscopy, or a history of uterine cavity surgery or uterine malformation correction
* Subjects who require placement of an intrauterine device or administration of oral contraceptives or subcutaneous implants after the procedure
* Individuals with mental status or cognitive function abnormalities who are unable to cooperate with the treatment process
* Subjects who, in the opinion of the investigator, have potential risks or any other factors that may interfere with the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy can happened to female only.
Enrollment: 200 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The thickness of the endometrium | The 21st day after induced abortion surgery
  Measurement of endometrial thickness by B-ultrasound on the 21st day after induced abortion surgery
Cycle normalization rate | 21st day of the first post-operative menstrual cycle
  proportion of ovarian function recovery; blood sampling for estradiol and progesterone level check on the 21st day of the first post-operative menstrual cycle

SECONDARY OUTCOMES:
Duration of vaginal bleeding after surgery | The 21st day after induced abortion surgery
  number of days of vaginal bleeding after induced abortion surgery
menstrual flow volume | 21st day of the first post-operative menstrual cycle
  Amount of menstrual flow during the first menstrual cycle after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxiu Jiang, Ph.D, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No